CLINICAL TRIAL: NCT00567333
Title: Individualized Chiropractic and Integrative Care for Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern Health Sciences University (Other)
Collaborators: Health Resources and Services Administration (HRSA) (U.S. Federal Agency); Berman Center for Outcomes and Clinical Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R18HP07639; R18HP07639
Record Dates: First submitted 2007-12-03; First posted 2007-12-04 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2015-05

CONDITIONS: Sub-Acute and Chronic Low Back Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Other)
  Interventions: Other: Chiropractic care
- 2 (Other)
  Interventions: Other: Multidisciplinary, integrative care

INTERVENTIONS:
Other: Chiropractic care — A combination of professional therapies with the scope of practice, including spinal manipulation therapy, spinal mobilization, stretching and strengthening exercises, and self-care education.
  Arms: 1
Other: Multidisciplinary, integrative care — A combination of therapies which may include acupuncture/Oriental medicine, chiropractic, cognitive behavioral therapy, exercise therapy, medicine, self-care information, and massage therapy.
  Arms: 2

SUMMARY:
This study proposes to compare two innovative treatment approaches for LBP, both of which focus on delivering individualized care through evidence-based, clinical care pathways.

The primary aim of the project is to determine the relative clinical efficacy of 1) chiropractic care and 2) multidisciplinary, integrative care in 200 patients with sub-acute or chronic LBP, in both the short-term (after 12 weeks) and long-term (after 52 weeks). The primary outcome measure in this study is patient-rated back pain.

Chiropractic care will include therapies within the professional scope of practice. Integrative, multidisciplinary care will include chiropractic, massage therapy, traditional Chinese medicine (including acupuncture), medication, cognitive behavioral therapy, exercise, and patient education.

Secondary aims are to assess between group differences in frequency of symptoms, disability, fear avoidance behavior, self efficacy, general health, improvement, patient satisfaction, work loss, medication use, lumbar dynamic motion, and torso muscle endurance. Patients' and providers' perceptions of treatment will be described using qualitative methods and cost-effectiveness and cost utility will be assessed in the short- and long-term.

This innovative study is an exciting collaboration between an experienced and established team of chiropractic, conventional, and CAM professionals dedicated to advancing the care of pervasive and costly LBP conditions. This trial will provide new and important information for all health care providers and LBP patients, informing decision making and improving care delivery systems.

ELIGIBILITY:
Inclusion Criteria:

* Mechanical LBP classified as 1, 2, 3, or 4 using Quebec Task Force (QTF) classification.70 (This includes back pain, stiffness or tenderness with or without musculoskeletal and neurological signs).
* LBP localized to posterior aspect of body, below the costal margin and above the inferior gluteal folds.
* Pain level > 3 on 0 to 10 scale
* Current LBP episode > 6 weeks duration
* 18 years of age and older
* Stable prescription medication plan (No changes in prescription medications that affect musculoskeletal pain in the previous month.)

Exclusion Criteria:

* Ongoing treatment for LBP by other non-study providers
* Progressive neurological deficits or cauda equina syndrome
* QTF classifications 5 (spinal instability or fracture) and 11 (other diagnoses including visceral diseases, compression fractures, metastases). These are serious conditions not amenable to the conservative treatments proposed.
* QTF 7 (Spinal stenosis syndrome characterized by pain and/or paresthesias in one or both legs aggravated by walking).
* Uncontrolled hypertension or metabolic disease
* Blood clotting disorders
* Severe osteoporosis
* Inflammatory or destructive tissue changes of the spine
* Patients with surgical lumbar spine fusion or patients with multiple incidents of lumbar surgery. This is a subgroup of LBP patients which generally have a poorer prognosis.
* Pregnant or nursing women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2007-06; Primary Completion 2010-10 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Patient-rated back pain. | Short term: 12 weeks, Long term: 52 weeks

SECONDARY OUTCOMES:
Frequency of Symptoms | 12 and 52 weeks
Low Back Disability | 12 and 52 weeks
Fear Avoidance | 12 and 52 weeks
Self-Efficacy | 12 and 52 weeks
General Health Status | 12 and 52 weeks
Improvement | 12 and 52 weeks
Patient Satisfaction | 12 and 52 weeks
Work Loss | 12 and 52 weeks
Medication Use | 12 and 52 weeks
Objective biomechanical measurements: Lumbar Dynamic Motion and Torso Muscle Endurance. | Short term: 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Gert Bronfort, DC, PhD, Principal Investigator — Northwestern Health Sciences University
Locations (1):
- Northwestern Health Sciences University, Bloomington, Minnesota, United States

REFERENCES:
- [Derived] Bronfort G, Maiers M, Schulz C, Leininger B, Westrom K, Angstman G, Evans R. Multidisciplinary integrative care versus chiropractic care for low back pain: a randomized clinical trial. Chiropr Man Therap. 2022 Mar 1;30(1):10. doi: 10.1186/s12998-022-00419-3. PMID 35232482
- [Derived] Maiers MJ, Westrom KK, Legendre CG, Bronfort G. Integrative care for the management of low back pain: use of a clinical care pathway. BMC Health Serv Res. 2010 Oct 29;10:298. doi: 10.1186/1472-6963-10-298. PMID 21034483
- [Derived] Westrom KK, Maiers MJ, Evans RL, Bronfort G. Individualized chiropractic and integrative care for low back pain: the design of a randomized clinical trial using a mixed-methods approach. Trials. 2010 Mar 8;11:24. doi: 10.1186/1745-6215-11-24. PMID 20210996